CLINICAL TRIAL: NCT03813199
Title: Phase IIa Randomized, Double Blind, Placebo Controlled, Multiple Dose Study on ABX464 in Combination With Methotrexate (MTX), in Patients With Moderate to Severe Active Rheumatoid Arthritis Who Have Inadequate Response to MTX or/and to Anti-Tnfα, or Intolerance to Anti-Tnfα
Brief Title: Study of Two Doses of ABX464 in Participants With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABX464-301
Record Dates: First submitted 2019-01-15; First posted 2019-01-23 (Actual); Results first posted 2022-04-07 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ABX464; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABX464 50mg + methotrexate (Experimental): Participants will receive one capsule of 50mg ABX464 plus one capsule of matching placebo once daily for 12 weeks
  + methotrexate
  Interventions: Drug: ABX464 50mg; Drug: Matching Placebo; Drug: Methotrexate
- ABX464 100mg + methotrexate (Experimental): Participants will receive two capsules of 50mg ABX464 once daily for 12 weeks
  + methotrexate
  Interventions: Drug: ABX464 100mg; Drug: Methotrexate
- Placebo + methotrexate (Placebo Comparator): Participants will receive two capsules of matching placebo once daily for 12 weeks
  + methotrexate
  Interventions: Drug: Matching Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: ABX464 50mg — ABX464 is a new anti-inflammatory drug
  Other Names: obefazimod 50mg
  Arms: ABX464 50mg + methotrexate
Drug: Matching Placebo — placebo matching with ABX464
  Other Names: Placebo
  Arms: ABX464 50mg + methotrexate; Placebo + methotrexate
Drug: ABX464 100mg — ABX464 is a new anti-inflammatory drug
  Other Names: obefazimod 100mg
  Arms: ABX464 100mg + methotrexate
Drug: Methotrexate — MTX ≥ 10 mg/week will be given at previous dose regimen kept stable throughout the study
  Other Names: MTX

SUMMARY:
This Phase IIa study aims at investigating the safety and tolerability of 2 dose-levels of ABX464 administered daily in combination with methotrexate (MTX) in patients with moderate to severe active Rheumatoid Arthritis (RA) who had an inadequate response to MTX or/and to one or more anti- tumor necrosis factor alpha (TNFα) therapies.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter study. The study will consist of 3 phases: a screening phase, a treatment phase, and a follow-up phase.

Approximately 60 participants with active Rheumatoid Arthritis will be randomly assigned to receive placebo, 50mg ABX464 or 100mg ABX464 during the treatment phase.

The maximum period of active treatment will be 12 weeks. The maximum duration of study participation will be 17 weeks.

Participant safety will be monitored throughout the study. In addition, several experimental and clinical endpoints will be assessed to obtain information on preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a confirmed and documented diagnosis of adult-onset rheumatoid arthritis, for at least 12 weeks, according to the revised 2010 American College of Rheumatology- European League Against Rheumatism (ACR-EULAR) classification criteria, including at least one positive criteria among the following: Rheumatoid Factor (RF), Anti-Citrullinated Peptide Antibody (ACPA) or bone erosion;
* Swollen joint count (SJC) of ≥ 4 (28-joint count) and tender joint count (TJC) ≥4 (28-joint count) at screening;
* Patient with a moderate to severe disease activity score Disease Activity Score (28 joints) C-Reactive Protein [DAS28 CRP] ≥ 3.2 and C-reactive Protein (CRP) ≥ 5 mg/L (≥ 4.76 nmol)/L) at screening;
* Patient who had an inadequate response (IR), or failed either methotrexate (MTX) or/and anti- Tumor Necrosis Factor alpha (TNFα) therapy (both administered for at least 12 weeks before IR) or were intolerant to anti- TNFα therapy.

Exclusion Criteria:

* Patient with a known positive anti-double stranded deoxyribonucleic acid (DNA [anti-dsDNA]) and confirmed diagnosis of systemic lupus erythematosus (SLE);
* Patient with known active infections at screening such as CytoMegaloVirus (CMV), herpes virus and/or recent infectious hospitalization;
* Acute, chronic or history of clinically relevant pulmonary, cardiovascular, hepatic, pancreatic or renal functional abnormality, encephalopathy, neuropathy or unstable Central Nervous System (CNS) pathology such as seizure disorder, angina or cardiac arrhythmias, active malignancy or any other clinically significant medical problems as determined by physical examination and/or laboratory screening tests and/or medical history;
* Acute, chronic or history of immunodeficiency or other autoimmune disease;
* Patient previously treated with any non-anti-TNF biological Disease-Modifying AntiRheumatic Drugs (bDMARDs), and targeted DMARDs (tDMARDS) prior to baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul GINESTE, PharmD, Study Director — Abivax S.A.
Locations (24):
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - ZNA Jan Palfijn, Merksem
- Czechia (2):
  - Fakultni Tomayerova nemocnice, Prague
  - Revmatologicky ustav, Prague
- France (8):
  - CHU de Brest - Hôpital Cavale Blanche, Brest
  - CHD Vendée, La Roche-sur-Yon
  - CHU de Montpellier - Lapeyronie, Montpellier
  - GHR Mulhouse Sud-Alsace, Mulhouse
  - CHU de Nice - Hôpital Pasteur, Nice
  - CHR d'Orléans, Orléans
  - APHP - Hôpital Salpétrière, Paris
  - CHU de Tours - Hôpital Trousseau, Tours
- Hungary (3):
  - Complex Medical Centre - Déli Klinika, Budapest
  - CRU Hungary Ltd., Miskolc
  - CMed Rehabilitációs és Diagnosztikai Központ, Székesfehérvár
- Poland (7):
  - ClinicMed Daniluk, Nowak Sp. J., Bialystok
  - Pratia MCM, Krakow
  - Zespół Poradni Specjalistycznych REUMED, Lublin
  - NZOZ Lecznica MAK-MED S.C., Nadarzyn
  - Medyczne Centrum Hetmańska, Poznan
  - National Institute of Geriatrics, Warsaw
  - RHEUMA MEDICUS Zakład Opieki Zdrowotnej, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daien C, Krogulec M, Gineste P, Steens JM, Desroys du Roure L, Biguenet S, Scherrer D, Santo J, Ehrlich H, Durez P. Safety and efficacy of the miR-124 upregulator ABX464 (obefazimod, 50 and 100 mg per day) in patients with active rheumatoid arthritis and inadequate response to methotrexate and/or anti-TNFalpha therapy: a placebo-controlled phase II study. Ann Rheum Dis. 2022 Jul 12;81(8):1076-1084. doi: 10.1136/annrheumdis-2022-222228. PMID 35641124

RESULTS

PARTICIPANT FLOW:
Groups:
- ABX464 50mg + Methotrexate: Participants will receive one capsule of 50mg ABX464 plus one capsule of matching placebo once daily for 12 weeks
  + methotrexate
  ABX464 50mg: ABX464 is a new anti-inflammatory drug
  Matching Placebo: placebo matching with ABX464
  Methotrexate: MTX ≥ 10 mg/week will be given at previous dose regimen kept stable throughout the study
- ABX464 100mg + Methotrexate: Participants will receive two capsules of 50mg ABX464 once daily for 12 weeks
  + methotrexate
  ABX464 100mg: ABX464 is a new anti-inflammatory drug
  Methotrexate: MTX ≥ 10 mg/week will be given at previous dose regimen kept stable throughout the study
- Placebo + Methotrexate: Participants will receive two capsules of matching placebo once daily for 12 weeks
  + methotrexate
  Matching Placebo: placebo matching with ABX464
  Methotrexate: MTX ≥ 10 mg/week will be given at previous dose regimen kept stable throughout the study
Period: Overall Study
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Started | 21 | 19 | 20
Completed | 18 | 6 | 19
Not Completed | 3 | 13 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate | Total
Number analyzed (Participants) | 21 | 19 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.4) | 54.4 (10.6) | 58.6 (11.0) | 57.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 11 | 37
  Male | 6 | 8 | 9 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events in the ABX464 Treated Patients Versus Placebo
Description: TEAE definition is undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment
Time Frame: through study completion, an average of 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
Participants | 18 | 18 | 14

2. Secondary Outcome: Number of Patients Achieving ACR20 Response
Description: The categorical American College of Rheumatology 20% (ACR20) response is a validated index of rheumatoid arthritis disease activity, defined by the number of patients who achieved at least 20% improvement in the ACR response.
Time Frame: at Week 12
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
Participants | 9 | 3 | 4

3. Secondary Outcome: Number of Patients Achieving ACR20/50/70 Response
Description: Number of patients who achieved at least 20%, 50% or 70% improvement in the American College of Rheumatology (ACR) response.
Time Frame: Week 12
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
Participants
  ACR20 response | 9 | 3 | 4
  ACR50 response | 5 | 2 | 1
  ACR70 response | 4 | 1 | 1

4. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP)
Description: Change from baseline in C-reactive protein (CRP) at Week 12
Time Frame: Week 12
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
mg/L | -4.31 (28.83) | 0.62 (4.89) | -0.65 (18.74)

5. Secondary Outcome: Number of Patients Achieving DAS28-CRP Response
Description: Number of patients achieving categorical Disease Activity Score (DAS) DAS28-C-Reactive Protein (CRP) [DAS28-CRP] response will be measured as moderate/good European League Against Rheumatism (EULAR) response
Time Frame: Week 12
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
Participants | 14 | 6 | 8

6. Secondary Outcome: Change From Baseline in Disease Activity Scores (DAS-CRP) (28 Joints) [DAS28]
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. The DAS28 assessment include 28 tender and swollen joint counts (TJC and SJC), acute phase reactant (CRP ), and patient's global assessment of disease activity (PtGA).
  DAS28-CRP = 0.56 √ (TJC28) + 0.28 √ (SJC28) + 0.36 Ln [CRP(mg/L)+1] + 0.014 PtGA(VAS100mm) + 0.96 Score scale range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Week 12
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
score on a scale | -1.41 (1.45) | -0.72 (1.13) | -0.60 (0.98)

7. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: Change from baseline in erythrocyte sedimentation rate (ESR) at Week 12
Time Frame: Week 12
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
mm/h | -2.6 (19.3) | -0.3 (6.8) | -2.7 (16.6)

8. Secondary Outcome: Number of Patients Achieving Disease Activity Score (DAS) DAS28-Erythrocyte Sedimentation Rate (ESR) [DAS28-ESR] Remission
Description: Number of patients achieving Disease Activity Score (DAS) DAS28-Erythrocyte Sedimentation Rate (ESR) [DAS28-ESR]remission, which is defined as DAS2-ESR < 2.6
Time Frame: Week 12
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
Participants | 2 | 0 | 0

9. Secondary Outcome: Change From Baseline in Disease Activtiy Score (DAS)28-Erythrocyte Sedimentation Rate (ESR)
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. The DAS28 assessment include 28 tender and swollen joint counts (TJC and SJC), acute phase reactant (ESR), and patient's global assessment of disease activity (PtGA).
  DAS28-ESR = 0.56 √ (TJC28) + 0.28 √ (SJC28) + 0.70 Ln [ESR(mm/h)] + 0.014 PtGA(VAS100mm) Score scale range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
  change from baseline at weeks 12: the bigger negative score shows a bigger improvment
Time Frame: 12 weeks
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
mm/h | -1.43 (1.39) | -0.74 (1.11) | -0.59 (1.00)

10. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index Score (SDAI)
Description: SDAI is a validated index of rheumatoid arthritis disease activity. The SDAI calculation is based on 28 tender and swollen joint counts, C-Reactive Protein (CRP), patient's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PrGA).
  SDAI score= tender28 + swollen28 + CRP + (PtGA/10) + (PrGA/10). A moderate activity is defined by a SDAI score >11 to 26 included. A high activity is defined by a SDAI score >26. Change from Baseline: the higher negative number shows a bigger improvment
Time Frame: Week 12
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
score on a scale | -20.21 (33.27) | -9.37 (14.44) | -7.58 (22.69)

11. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index Score (CDAI)
Description: CDAI is a validated index of rheumatoid arthritis disease activity. The CDAI calculation is based on 28 tender and swollen joint counts, patient's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PrGA).
  CDAI score= tender28 + swollen28 + (PtGA/10) + (PrGA/10). A moderate activity is defined by a CDAI score >10 to 22 included. A high activity is defined by a CDAI score >22. Change from Baseline: the higher negative number shows a bigger improvment
Time Frame: Week 12
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
score on a scale | -15.89 (13.29) | -9.99 (15.85) | -6.93 (10.13)

12. Secondary Outcome: Number of Patients Achieving Low Disease Activity (LDA)
Description: Number of patients achieving a Low Disease Activity (LDA) which is defined as DAS28-ESR <=3.2
Time Frame: Week 12
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
Participants | 4 | 2 | 2

13. Secondary Outcome: Number of Patients Achieving Simplified Disease Activity Score (SDAI) Remission
Description: Number of patients achieving Simplified Disease Activity Score (SDAI) remission, which is considered achieved if the SDAI score ≤ 3.3
Time Frame: Week 12
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
Participants | 1 | 0 | 0

14. Secondary Outcome: Number of Patients Achieving Clinical Disease Activity (CDAI) Remission
Description: Number of patients achieving Clinical Disease Activity (CDAI) remission, which is considered achieved if the CDAI score ≤ 2.8
Time Frame: Week 12
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
Participants | 3 | 0 | 0

15. Secondary Outcome: Number of Patients Achieving American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Boolean Remission
Description: The ACR/EULAR boolean-based remission is a validated criteria based on: Tender/painful Joint Count (28), Swollen Joint Count (28), C-Reactive Protein, patient global assessment of disease, All ≤ 1
Time Frame: Week 12
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
Participants | 1 | 0 | 0

16. Secondary Outcome: Change From Baseline in Tender/Painful Joint Count (TJC28)
Description: Change from Baseline in Tender/painful joint count based on 28-joint assessment (TJC28) at Week 12 TJC28 score range from 0 to 28 Change from Baseline: the higher the negative number is, the better improvment is
Time Frame: 12 weeks
Population: intent to treat
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
joints | -6.8 (6.4) | -4.1 (6.6) | -2.9 (3.8)

17. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC)
Description: Change from Baseline in Swollen joint count based on 28-joint assessment (SJC28) at Week 12 SJC28 score range from 0 to 28 Change from Baseline: the higher the negative number is, the better improvment is
Time Frame: 12 weeks
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
joints | -4.4 (4.2) | -3.2 (5.3) | -2.1 (4.2)

18. Secondary Outcome: Change From Baseline in Pain Visual Analog Scale
Description: Change from Baseline in Pain Visual Analog Scale (Pain-VAS) at week 12 The VAS range from 0 to 10 cm (the higher, the more painful) A bigger negative change from baseline shows a bigger improvment
Time Frame: 12 weeks
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
units on a scale | -2.63 (2.43) | -0.89 (1.97) | -0.78 (2.36)

19. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease (PtGA)
Description: Change from Baseline in Patient Global Assessment of Disease (PtGA) . This is a patient's self assessment of overall RA disease activity on a scale 1-10 where 10 is maximal activity The change from baseline: a bigger negative number shows a bigger improvment
Time Frame: 12 weeks
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
units on a scale | -1.44 (1.92) | -0.89 (1.93) | -0.36 (2.16)

20. Secondary Outcome: Change From Baseline in Investigator Global Assessment of Disease (PrGA)
Description: Change from Baseline in Investigator global assessment of disease (PrGA): investigator's assessment of overall RA disease activity on a scale 1-10 where 10 is maximal activity The change from baseline: the higher negative number shows a better improvement
Time Frame: 12 weeks
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
units on a scale | -3.26 (2.7) | -1.89 (2.95) | -1.63 (2.38)

21. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: Change from Baseline in Health Assessment questionnaire disability index (HAQ-DI) at Week 12 There are 8 sections in this questionnaire: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section, i.e. if one question is scored 1 and another 2, then the score for the section is 2. In addition, if an aide or device is used or if help is required from another individual, then the minimum score for that section is 2.
  The 8 scores of the 8 sections are summed and divided by the number of section answered.
  This gives a score range from 0 to 3 (the bigger the worst activity). The change from Baseline: the bigger negative number shows a bigger improvment
Time Frame: 12 weeks
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 21 | 19 | 20
units on a scale | -0.4345 (0.6182) | -0.1053 (0.3443) | -0.1813 (0.4824)

ADVERSE EVENTS:
Time Frame: 15 weeks
Arm/Group | ABX464 50mg + Methotrexate | ABX464 100mg + Methotrexate | Placebo + Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/19 | 1/20
Other Adverse Events (participants affected / at risk) | 15/21 | 17/19 | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 50mg + Methotrexate (N=21) | ABX464 100mg + Methotrexate (N=19) | Placebo + Methotrexate (N=20)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — atrial fibrillation reactive to hypokalemia secondary to diarrhea in the context of study drug treatment
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 50mg + Methotrexate (N=21) | ABX464 100mg + Methotrexate (N=19) | Placebo + Methotrexate (N=20)
Headache (Nervous system disorders) | 8 (19) | 10 (16) | 4 (6)
nausea (Gastrointestinal disorders) | 3 (4) | 9 (12) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 7 (11) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 4 (10) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT03813199/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT03813199/SAP_001.pdf